CLINICAL TRIAL: NCT01840046
Title: Evaluation of the Efficacy and Tolerability of Treatment With Interleukin-2 in Severe Alopecia Areata Resistant to Conventional Systemic Treatment
Brief Title: Evaluation of the Efficacy and Tolerability of Treatment With Interleukin-2 in Severe and Resistant Alopecia Areata
Acronym: IL2
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-PP-05
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2013-03

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interleukin 2 (Experimental): The patient will receive 4 cycles of recombinant interleukin 2 (aldesleukin, Proleukin ®) subcutaneously according to the following dosing schedule:
  5 to 7 days (Monday to Friday) in weeks 1, 3, 6 and 9.
  The dosage is as follows:
  S1: 1.5 mille-International unit (MIU) / day D1 to D5, S3, S6 and S9: 3 mille-International unit /Jour D1 to D5.
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — The patient will receive 4 cycles of recombinant interleukin 2 (aldesleukin, Proleukin ®) subcutaneously according to the following dosing schedule:
  5 to 7 days (Monday to Friday) in weeks 1, 3, 6 and 9.
  The dosage is as follows:
  S1: 1.5 mille-International unit / day (D1 to D5), S3, S6 and S9: 3 mille-International unit /Jour (D1 to D5).

SUMMARY:
Alopecia areata is an autoimmune disease associated with infiltration of cluster of differentiation 4(CD4 +) and cluster of differentiation 8 (CD8) + cells around the hair follicles. One of the therapeutic approaches of inflammatory diseases such as alopecia areata is the induction of tolerance. This tolerance induction can be obtained by stimulating regulatory T cells (Treg). The low-dose interleukin-2 plays a central role in the development, expansion, regulation and survival of regulatory T cells CD4 + cluster of differentiation 25 (CD25) + forkhead box protein 3 (FoxP3). Recently, recombinant interleukin 2 (IL2-R) with low dose showed very promising results in two inflammatory disease (GVHD vasculitis and cryoglobulinemia secondary to hepatitis C): clinical efficacy, increased population Treg in the blood and an excellent safety profile. We hypothesized that administration of IL2-R in patients with severe alopecia areata might allow regrowth via activation of Treg and thus induce regrowth of the air.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, 60 ≤ years.
* Male or female
* Clinical diagnosis of alopecia areata,
* Severe alopecia areata (> 50% of the surface of the scalp reached)
* Alopecia areata resistant to at least one systemic therapy: phototherapy (UVB or PUVA), methotrexate or corticosteroids
* Signature of the informed consent and authorization of the right image
* Effective contraception will be maintained for the duration of the study.
* Affiliation to the Social Security

Exclusion Criteria:

* Pregnancy or refusal of contraception in women of childbearing age,
* Refusal of contraception for men
* Local treatment (corticosteroids, minoxidil) or systemic (oral corticosteroids, methotrexate or other immunosuppressive agents) for less than 2 months,
* Cancer or autoimmune disease or in remission evolutionary
* Excessive alcohol intake (more than 3 glasses of wine a day or a drink per day)
* HIV, hepatitis C virus, hepatitis B virus
* Patient with renal and / or hepatic impairment,
* Patient with shingles, chickenpox, herpes, tuberculosis, an infectious disease scalable, respiratory failure ...
* Vulnerable person (anyone younger, adults under guardianship, deprived of liberty)
* Indication against treatment with IL2-R
* Presenting an indication against the Proleukin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of patients who obtained an improvement of at least 90% of the score validated severity score in alopecia areata in 2 months. | 2 months
  Number of patients who obtained an improvement of at least 90% of SALT (SALT 90) validated severity score in alopecia areata in 2 months.

SECONDARY OUTCOMES:
Evaluation of the quality of life | 2 months
  Number of patients who obtained an improvement of at least 50% of score (SALT 90) validated severity score in alopecia areata in 2 months.
  Assess the partial response rate. Evaluation of the effects of treatment on body hair and nail achieving.
  Overall assessment by an independent investigator to regrow after treatment (Physician global assessment):
  Evaluation of the quality of life before and at the end of treatment. Overall assessment by the patient (patient global assessment) of regrowth. Overall tolerability of treatment. Study population effects of IL2-R on the population of Treg cells in the blood. The effects of IL-2 on the inflammatory infiltrate and the distribution of regulatory T cells in the skin.

CONTACTS AND LOCATIONS:
Overall Officials: PASSERON Thierry, PhD, Principal Investigator — CHU de Nice - Hôpital de l'Archet - Dermatology
Locations (1):
- CHU de Nice - Hôpital Archet, Nice, Alpes-Maritimes, France

REFERENCES:
- [Derived] Castela E, Le Duff F, Butori C, Ticchioni M, Hofman P, Bahadoran P, Lacour JP, Passeron T. Effects of low-dose recombinant interleukin 2 to promote T-regulatory cells in alopecia areata. JAMA Dermatol. 2014 Jul;150(7):748-51. doi: 10.1001/jamadermatol.2014.504. PMID 24872229